CLINICAL TRIAL: NCT01864265
Title: Prediction of Response to Certolizumab Pegol Treatment by Functional MRI of the Brain. A Multi-center, Randomized Double-blind Controlled Study Prediction of Response to Certolizumab-Pegol in RA (PreCePRA)
Brief Title: Prediction of Response to Certolizumab Pegol Treatment by Functional MRI of the Brain
Acronym: PreCePRA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PreCePRA
Record Dates: First submitted 2013-05-21; First posted 2013-05-29 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; functional MRI; Prediction of Response; Certolizumab Pegol
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Certolizumab Pegol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Certolizumab Pegol (Active Comparator)
  Interventions: Drug: Certolizumab Pegol; Drug: Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Certolizumab Pegol; Drug: Placebo

INTERVENTIONS:
Drug: Certolizumab Pegol — Certolizumab Pegol (Cimzia®) is an engineered, humanized antibody-Fab'-fragment with specificity for human TNF-α, that is conjugated to polyethylene glycol (PEG). Certolizumab Pegol (Cimzia®) is a humanized antibody-Fab'-fragment that is produced in Escherichia coli and subsequently PEGylated to prolong its circulating half-time to be similar to that of an intact mAB. Certolizumab Pegol has a high affinity for TNF α with a Kd90pM and is an effective TNF α inhibitor. Certolizumab pegol does not neutralize TNFß (lymphotoxin), a related cytokine, and does not activate complement or kill cells via antibody-dependent cellular toxicity.
  Other Names: Cimzia
Drug: Placebo — Placebo will be administered according to the label of the biological

SUMMARY:
By using functional MRI the investigators have recently shown that TNFi elicit rapid changes in brain function linked to the perception of RA [5]. Functional MRI represents a method allowing detecting tiny changes in neuronal activity by measuring alterations of blood flow in the context of neuronal activation. TNFi rapidly reversed the widespread activation of brain centers involved in pain such as the thalamus and the somatosensoric cortex, as well as those involved in the control, of mood and emotions such as the limbic system. Moreover, as small phase I study with 10 patients with RA showed that high brain activity detected in the functional MRI predicts clinical response to Certolizumab Pegol after 1 month, suggesting the central nervous system activity may be used as a tool to predict response to TNFi [8]. The rationale of this study is to test whether response to TNFi can be predicted by using functional MRI.

DETAILED DESCRIPTION:
Randomized double-blinded controlled multi-centre, study over 12 weeks, followed by a 12 weeks single blinded multicenter trial in 156 patients with RA with inadequate response to DMARD therapy. The study is composed of 3 arms with a 1:1:1 randomization at baseline: High functional MRI/400mg Certolizumab Pegol on week 0,2 and 4 followed by Certolizumab Pegol 200mg every two weeks for a total of 24 weeks; low functional MRI/400mg Certolizumab Pegol on week 0,2 and 4 followed by Certolizumab Pegol 200mg every two weeks for a total of 24 weeks with the possibility of early escape at week 12.

Patients who did not respond sufficiently according to EULAR response criteria (DAS28 reduction ≥ 1.2) to Certolizumab-Pegol (Treatment Arm A and Arm B) after 12 weeks will be off-Study and treated according to local guidelines.

Patients in the Placebo group with an EULAR response ≥ 1.2 reaching remission (DAS28 ≤ 2.6) will also be off study and treated according to the local guidelines or will be followed while they are in clinical remission. Patients with an EULAR response (DAS28 reduction ≥ 1.2) but not fulfilling the clinical remission criteria (DAS28 ≤ 2.6) will receive Certolizumab Pegol in week 12,14 and 16 with Certolizumab Pegol 400mg s.c. followed by s.c.injection of 200mg Certolizumab Pegol every two weeks till week 24.

In the situation that in one group sufficient patients will be randomized, fMRI done at screening, needs to be analyzed first to ensure that no further patient will be randomized with the randomization to the closed group. A blinded person, not involved either in the analysation of the fMRI nor in the treatment of the patients or the clinical assessments, will be responsible for the randomization list. If the next number on the randomization list represent the number of the closed group, the patient is not eligible for the study and will be treated according to local guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Understands and voluntarily signs an informed consent form
* Male or female, aged ≥ 18 years at time of consent
* Must be able to adhere to the study visit schedule and other protocol requirements
* Must satisfy the 2010 ACR/EULAR classification criteria for rheumatoid arthritis plus a disease duration of at least 6 months.
* Must have active RA with a DAS28 ≥3.2
* Must be RF and/or ACPA positive
* ≥ 3 swollen and/or tender joints of the hands
* At screening- visit patients should have been treated without alterations of therapy for at least three months with DMARDS (i.e. Methotrexate) with or without concomitant use of steroids).
* Glucocorticoids treatment up to 10mg prednisolone per day will be allowed at study entry.

  . Exclusion Criteria:
* Individuals not able to understand and follow study protocol and not able to voluntarily sign informed consent
* Individuals not willing to follow study protocol and sign informed consent
* Individuals with claustrophobia, tattoos containing metal, magnetic endoprostheses, surgery on bone in between a time interval < 3 months.
* Patients treated before with any biological or small molecule or medication under investigation for the treatment of RA.
* Patients with serious or chronic infections within the previous 3 months
* Opportunistic infections within the 6 months before screening
* Cancer within the 5 years before screening (with the exception of treated and cured squamous or basal cell carcinoma of the skin)
* History of severe congestive heart failure
* Current signs or symptoms of severe, progressive, or uncontrolled renal, hepatic, hematologic, gastrointestinal (a.e.diverticulitis), endocrine, pulmonary, cardiac, neurologic or cerebral disease
* Transplanted organ (with the exception of corneal transplantation done more than 3 months before screening)
* Evidence of active tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2013-07; Primary Completion 2019-06-30 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Reaching low disease activity | 6 months
  Proportion of patients who reach low disease activity according to the DAS28 (DAS28 < 3.2) during the first 12 weeks of study participation according their screening CNS activity measured by functional MRI.

SECONDARY OUTCOMES:
Remission | 6 months
  Proportion of subjects in each treatment group reaching remission (defined as DAS28 < 2.6) after 1, 12 and 24 weeks
Quality of Life | 6 months
  HAQ of zero after 12 and 24 weeks to baseline
SF36 | 6 months
  Mean and median SF-36 after 1, 12 and 24 weeks
MRI | 6 months
  Proportion of subjects in each treatment group with normal functional MRI after screening, week 12 and 24 weeks
Normal fMRI | 6 months
  Proportion of subjects in each treatment group with normal functional MRI after screening, 12 and 24 weeks
Ultrasound score | 6 months
  Mean and median ultrasound synovitis score after 1, 12 and 24 weeks
Bold signal | 6 months
  Mean and median ultrasound synovitis score after 1, 12 and 24 weeks
Adverse events | 6 months
  Type, frequency, severity and relationship of adverse events, serious adverse events or suspected unexpected serious adverse reactions to drugs used in this study
Number of patients who discontinue Certolizumab-Pegol | 6 months
  Number of subjects who prematurely discontinue Certolizumab-Pegol due to any adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Rech, MD, Principal Investigator — University of Erlangen-Nuremberg, Department of Internal Medicine 3, Rheumatology & Immunology; Georg Schett, MD, Prof., Study Director — University of Erlangen-Nuremberg, Department of Internal Medicine 3, Rheumatology & Immunology
Locations (6):
- Germany (4):
  - Charité - Universitätsmedizin Berlin; Campus Charité Mitte Klinik für Rheumatologie und klinische Immunologie Studienambulanz, Berlin
  - University of Erlangen-Nuremberg, Department of Internal Medicine 3, Rheumatology & Immunology, Erlangen
  - Medizinische Universitätsklinik Freiburg Abteilung Rheumatologie und Klinische Immunologie, Freiburg im Breisgau
  - Universitätsklinikum Leipzig AÖR Department Innere Medizin Sektion Rheumatologie, Leipzig
- Hospitais da Universidade (SRHUC) Reumatologia, Coimbra, Portugal
- Belgrade University School of Medicine Director of the Institute Institute of Rheumatology, Belgrade, Serbia

REFERENCES:
- [Derived] Hess A, Tascilar K, Schenker HM, Konerth L, Schonau V, Sergeeva M, Kreitz S, Prade J, Strobelt S, Selvakumar M, Kleyer A, Englbrecht M, Hueber AJ, Zaiss MM, Feist E, Burmester GR, Voll RE, Finzel S, Baerwald C, Rosch J, Behrens F, Koehm M, da Silva JAP, Damjanov N, Dorfler A, Schett G, Rech J. Disease-associated brain activation predicts clinical response to TNF inhibition in rheumatoid arthritis (PreCePra): a randomised, multicentre, double-blind, placebo-controlled phase 3 study. Lancet Rheumatol. 2025 Aug;7(8):e565-e575. doi: 10.1016/S2665-9913(25)00032-3. Epub 2025 Jun 23. PMID 40570879